CLINICAL TRIAL: NCT01212809
Title: A Prospective, Open Label, Randomized, Comparative, Split-Face Study Evaluating Reconstituted JUVÉDERM® Ultra Injectable Gel Versus COSMODERM® 1 Human Based Collagen Implant for the Treatment of Vertical Lip Rhytids and Radial Cheek Lines
Brief Title: Comparative Study of Reconstituted JUVÉDERM® Ultra vs COSMODERM® 1 for Lip and Cheek Lines, Folds or Wrinkles
Acronym: JUVE_COSMO_1
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Steven Fagien (Other)
Responsible Party: Sponsor-Investigator, Steven Fagien, Principal Investigator, Fagien, Steven, M.D., PA
Organization: Fagien, Steven, M.D., PA (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: JUVE_COSMO_1-10-01
Record Dates: First submitted 2010-09-29; First posted 2010-10-01 (Estimated); Last update posted 2011-09-12 (Estimated); Status verified 2011-09

CONDITIONS: Intrinsic Aging of Skin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Juvéderm Ultra (Active Comparator): Juvéderm Ultra injection
  Interventions: Device: Juvéderm Ultra
- Cosmoderm 1 (Active Comparator): Cosmoderm 1 injection
  Interventions: Device: Cosmoderm 1

INTERVENTIONS:
Device: Juvéderm Ultra — Split-face injection of Juvéderm Ultra into vertical lip rhytids and radial cheek lines on one side of face
  Other Names: Juvéderm Ultra injectable gel (crosslinked hyaluronic acid)
  Arms: Juvéderm Ultra
Device: Cosmoderm 1 — Split-face injection of Cosmoderm 1 into vertical lip rhytids and radial cheek lines on one side of face
  Other Names: Cosmoderm 1 human-based collagen implant
  Arms: Cosmoderm 1

SUMMARY:
This study is being done to evaluate the differences in the performance of two well known injectable dermal fillers commonly used for the cosmetic treatment of age lines above the lips and on the cheeks when compared to each other in the same patient. The products being tested are Juvéderm® Ultra and CosmoDerm® 1.

DETAILED DESCRIPTION:
This is a single center, prospective, open label, randomized, comparative, split-face study in adult females or males aged 25 to 70 years seeking treatment with reconstituted Juvéderm® Ultra and CosmoDerm® 1 human-based collagen implant for moderate to severe vertical lip rhytids and/or radial cheek lines.

ELIGIBILITY:
Inclusion Criteria:

* Adult females or males, aged 25 to 70 years;
* Subjects must be seeking treatment with Juvéderm Ultra and CosmoDerm 1 injections for vertical lip rhytids or radial cheek lines;
* Subjects must have one or more moderate to severe vertical lip rhytids and/or moderate to severe radial cheek lines based on the physician evaluator assessment (0-3 scale);
* Women must either be of non-childbearing potential (i.e., surgically sterilized or post-menopausal) or if of childbearing potential, must not be pregnant (as documented by a negative urine pregnancy test at the baseline examination) or lactating and must be practicing a medically acceptable method of birth control;
* Subjects must be willing and able to provide written informed consent;
* Subjects must be willing and able to follow the procedures outlined in this protocol.

Exclusion Criteria:

* Female subjects who are pregnant (positive urine pregnancy test) or who have an infant they are breast-feeding or who are of childbearing potential and not practicing a reliable method of birth control;
* Previous Botox treatment to the lower two-thirds of the face within the past 6 months for subjects who will have injections into their radial cheek lines. Note: this exclusion criterion does not apply to subjects who only will have injections into lip rhytids unless the previous Botox treatment was administered within the past 6 months to the upper lip region;
* Previous semipermanent injectable filler therapy to the mid-lower face within the past year or any prior history of permanent filler therapy injection to the mid-lower face;
* Prior cosmetic procedures (i.e., facelift, etc.) or visible scars that may affect evaluation of response and/or quality of photography in the opinion of the investigator;
* Known allergy or sensitivity to any of the treatment injections or their components, including known or suspected lidocaine hypersensitivity;
* Known severe allergies manifested by a history of anaphylaxis or history or presence of multiple severe allergies;
* Subjects with an infection at an injection site or systemic infection (in this case, postpone study entry until one week following recovery);
* Subjects requiring treatment with major anticoagulants (such as Coumadin) or antiplatelets (such as Plavix) during the study; low-dose aspirin treatment or antiinflammatory medication with potential anticoagulant or antiplatelet effect may be allowed at the investigator's discretion;
* Concurrent participation in an investigational drug or device study or participation within 30 days of study start;
* Subjects are not to undergo any additional cosmetic procedures during the study period;
* Subjects are not to change use of any facial products up to 6 months prior to enrollment and during study period;
* Subjects with a history of poor cooperation, non-compliance with medical treatment, or unreliability.

Ages: 25 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2010-09; Primary Completion 2011-04 (Actual); Study Completion 2011-06 (Actual)

PRIMARY OUTCOMES:
Global Assessment of Improvement by Physician Evaluator | 3 days, 2 and 6 weeks, 4 and 6 months
  Global Assessment of Improvement by Physician Evaluator, including Facial Photographs, Vertical Lip Rhytids and Radial Cheek Line Rating Scales

SECONDARY OUTCOMES:
Patient Efficacy, Pain, Adverse Event Assessments | 3 days, 2 and 6 weeks, 4 and 6 months
  * Facial Line Outcomes (FLO-11 version 1.0) Questionnaire - Patient
  * Self-Perception of Age (SPA version 2.0) measure - Patient
  * Global Assessment of Improvement - Patient
  * Self-Rated Pain Assessment Scale (0-10 point rating scale)
  * Treatment-emergent adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Steven Fagien, MD, Principal Investigator — Steven Fagien, MD, PA
Locations (1):
- Steven Fagien, MD, PA, Boca Raton, Florida, United States